CLINICAL TRIAL: NCT05553808
Title: A Phase II, Randomized, Open-label Platform Trial Utilizing a Master Protocol to Study Novel Regimens Versus Standard of Care Treatment in NSCLC Participants
Brief Title: Platform Trial of Novel Regimens Versus Standard of Care (SoC) in Participants With Non-small Cell Lung Cancer (NSCLC) - Sub-study 1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: iTeos Belgium SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 205801-001; 2018-001316-29 (EudraCT Number)
Record Dates: First submitted 2022-09-21; First posted 2022-09-23 (Actual); Results first posted 2023-01-19 (Actual); Last update posted 2023-01-19 (Actual); Status verified 2022-12

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms | interventions — Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Docetaxel (Active Comparator)
  Interventions: Drug: Docetaxel
- Feladilimab plus Docetaxel (Experimental)
  Interventions: Drug: Docetaxel; Drug: Feladilimab

INTERVENTIONS:
Drug: Docetaxel — Docetaxel was administered as IV infusion.
Drug: Feladilimab — Feladilimab was administered as IV infusion.
  Arms: Feladilimab plus Docetaxel

SUMMARY:
This study is a sub-study of the master protocol 205801 (NCT03739710). This sub study has assessed the clinical activity of novel regimen (Feladilimab plus Docetaxel) with SOC (Docetaxel) in participants with NSCLC.

ELIGIBILITY:
Inclusion Criteria:

* Participants capable of giving signed informed consent/assent.
* Male or female, aged 18 years or older at the time consent is obtained. Participants in Korea must be age 19 years or older at the time consent is obtained.
* Participants with histologically or cytologically confirmed diagnosis of NSCLC (squamous or non-squamous) and

  a) Documented disease progression based on radiographic imaging, during or after a maximum of 2 lines of systemic treatment for locally/regionally advanced recurrent, Stage IIIb/Stage IIIc/Stage IV or metastatic disease. Two components of treatment must have been received in the same line or as separate lines of therapy: i) No more than or less than 1 line of platinum-containing chemotherapy regimen, and ii) No more than or less than 1 line of Programmed cell death ligand 1 (PD[L]1) monoclonal antibody (mAb) containing regimen.

  b) Participants with known BRAF molecular alterations must have had disease progression after receiving the locally available SoC treatment for the molecular alteration.

  c) Participants who received prior anti-PD(L)1 therapy must fulfill the following requirements: i) Have achieved a CR, PR or SD and subsequently had disease progression (per RECIST 1.1 criteria) either on or after completing PD(L)1 therapy ii) Have not progressed or recurred within the first 12 weeks of PD(L)1 therapy, either clinically or per RECIST 1.1 criteria
* Measurable disease, presenting with at least 1 measurable lesion per RECIST 1.1.
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) score of 0 or 1.
* A tumor tissue sample obtained at any time from the initial diagnosis of NSCLC to time of study entry is mandatory. Although a fresh tumor tissue sample obtained during screening is preferred, archival tumor specimen is acceptable.
* Adequate organ function as defined in the protocol.
* A male participant must agree to use a highly effective contraception during the treatment period and for at least 120 days after the last dose of study treatment and refrain from donating sperm during this period.
* A female participant is eligible to participate if she is not pregnant, not breastfeeding, and at least 1 of the following conditions apply:

  i) Not a woman of childbearing potential (WOCBP) or ii) A WOCBP who agrees to follow the contraceptive guidance during the treatment period and for at least 120 days after the last dose of study treatment.
* Life expectancy of at least 12 weeks.

Exclusion Criteria:

* Participants who received prior treatment with the following therapies (calculation is based on date of last therapy to date of first dose of study treatment):

  1. Docetaxel at any time.
  2. Any of the investigational agents being tested in the current study.
  3. Systemic approved or investigational anticancer therapy within 30 days or 5 half-lives of the drug, whichever is shorter. At least 14 days must have elapsed between the last dose of prior anticancer agent and the first dose of study drug is administered.
  4. Prior radiation therapy: permissible if at least one non-irradiated measurable lesion is available for assessment per RECIST version 1.1 or if a solitary measurable lesion was irradiated, objective progression is documented. A wash out of at least 2 weeks before start of study drug for radiation of any intended use is required.
* Received greater than (>)2 prior lines of therapy for NSCLC, including participants with BRAF molecular alternations.
* Invasive malignancy or history of invasive malignancy other than disease under study within the last 2 years, except

  * Any other invasive malignancy for which the participant was definitively treated, has been disease-free for at least 2 years and in the opinion of the principal investigator and GlaxoSmithKline Medical Monitor will not affect the evaluation of the effects of the study treatment on the currently targeted malignancy, may be included in this clinical trial.
  * Curatively treated non-melanoma skin cancer or successfully treated in situ carcinoma.
* Carcinomatous meningitis (regardless of clinical status) and uncontrolled or symptomatic Central nervous system (CNS) metastases.
* Major surgery less than or equal to (<=) 28 days of first dose of study treatment.
* Autoimmune disease (current or history) or syndrome that required systemic treatment within the past 2 years. Replacement therapies which include physiological doses of corticosteroids for treatment of endocrinopathies (for example, adrenal insufficiency) are not considered systemic treatments.
* Receiving systemic steroids (>10 milligrams [mg]) oral prednisone or equivalent) or other immunosuppressive agents within 7 days prior to first dose of study treatment.
* Prior allogeneic/autologous bone marrow or solid organ transplantation.
* Receipt of any live vaccine within 30 days prior to first dose of study treatment.
* Toxicity from previous anticancer treatment that includes:

  1. Greater than or equal to (>=) Grade 3 toxicity considered related to prior immunotherapy and that led to treatment discontinuation.
  2. Toxicity related to prior treatment that has not resolved to <= Grade 1 (except alopecia, hearing loss, endocrinopathy managed with replacement therapy, and peripheral neuropathy which must be <= Grade 2).
* History (current and past) of idiopathic pulmonary fibrosis, pneumonitis (for past- pneumonitis exclusion only if steroids were required for treatment), interstitial lung disease, or organizing pneumonia.
* Recent history (within the past 6 months) of uncontrolled symptomatic ascites, pleural or pericardial effusions.
* Recent history (within the past 6 months) of gastrointestinal obstruction that required surgery, acute diverticulitis, inflammatory bowel disease, or intra-abdominal abscess.
* History or evidence of cardiac abnormalities within the 6 months prior to enrollment which include

  1. Serious, uncontrolled cardiac arrhythmia or clinically significant electrocardiogram abnormalities including second degree (Type II) or third degree atrioventricular block.
  2. Cardiomyopathy, myocardial infarction, acute coronary syndromes (including unstable angina pectoris), coronary angioplasty, stenting or bypass grafting.
  3. Symptomatic pericarditis.
* Current unstable liver or biliary disease per investigator assessment defined by the presence of ascites, encephalopathy, coagulopathy, hypo-albuminemia, esophageal or gastric varices, persistent jaundice, or cirrhosis.
* Active infection requiring systemic therapy <=7 days prior to first dose of study treatment.
* Participants with known human immunodeficiency virus infection.
* Participants with history of severe hypersensitivity to mAb or hypersensitivity to any of the study treatment(s) or their excipients.
* Participants requiring ongoing therapy with a medication that is a strong inhibitor or inducer of the cytochrome P 3A4 (CYP3A4) enzymes.
* Any serious and/or unstable pre-existing medical (aside from malignancy), psychiatric disorder, or other condition that could interfere with participant's safety, obtaining informed consent, or compliance to the study procedures in the opinion of the investigator.
* Pregnant or lactating female participants.
* Participant who is currently participating in or has participated in a study of an investigational device within 4 weeks prior to the first dose of study treatment.
* Participants with presence of hepatitis B surface antigen (HBsAg) at screening or within 3 months prior to first dose of study intervention.
* Participants with positive hepatitis C antibody test result at screening or within 3 months prior to first dose of study intervention.
* Participants with positive hepatitis C ribonucleic acid (RNA) test result at screening or within 3 months prior to first dose of study treatment.
* Receipt of transfusion of blood products (including platelets or red blood cells) or administration of colony-stimulating factors (including granulocyte colony stimulating factor [G-CSF], granulocyte-macrophage colony-stimulating factor, and recombinant erythropoietin) within 14 days before the first dose of study intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2019-01-24 (Actual); Primary Completion 2021-09-23 (Actual); Study Completion 2021-09-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (38):
- United States (3):
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Nashville, Tennessee
  - GSK Investigational Site, Dallas, Texas
- GSK Investigational Site, Toronto, Ontario, Canada
- France (5):
  - GSK Investigational Site, Bordeaux
  - GSK Investigational Site, Caen
  - GSK Investigational Site, Nantes
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Villejuif
- Germany (5):
  - GSK Investigational Site, Gauting, Bavaria
  - GSK Investigational Site, Immenhausen, Hesse
  - GSK Investigational Site, Leipzig, Saxony
  - GSK Investigational Site, Großhansdorf, Schleswig-Holstein
  - GSK Investigational Site, Berlin
- Italy (4):
  - GSK Investigational Site, Meldola (FC), Emilia-Romagna
  - GSK Investigational Site, Ravenna, Emilia-Romagna
  - GSK Investigational Site, Milan, Lombardy
  - GSK Investigational Site, Orbassano (TO), Piedmont
- GSK Investigational Site, Maastricht, Netherlands
- Poland (3):
  - GSK Investigational Site, Lodz
  - GSK Investigational Site, Poznan
  - GSK Investigational Site, Warsaw
- Romania (5):
  - GSK Investigational Site, Bucharest
  - GSK Investigational Site, Craiova
  - GSK Investigational Site, Floreşti
  - GSK Investigational Site, Otopeni
  - GSK Investigational Site, Timișoara
- Russia (2):
  - GSK Investigational Site, Chelyabinsk
  - GSK Investigational Site, Saint Petersburg
- South Korea (4):
  - GSK Investigational Site, Cheongju-si
  - GSK Investigational Site, Gyeonggi-do
  - GSK Investigational Site, Seongnam
  - GSK Investigational Site, Seoul
- Spain (4):
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Santander
  - GSK Investigational Site, Seville
- GSK Investigational Site, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to anonymized individual patient-level data (IPD) and related study documents of the eligible studies via the Data Sharing Portal. Details on GSK's data sharing criteria can be found at: https://www.gsk.com/en-gb/innovation/trials/data-transparency/
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk.com/en-gb/innovation/trials/data-transparency/

RESULTS

PARTICIPANT FLOW:
Groups:
- Docetaxel 75 mg/m^2: Participants with NSCLC were administered with Docetaxel 75 milligram per meter square (mg/m^2) monotherapy as intravenous (IV) infusion once every 3 weeks (Q3W).
- Feladilimab 80 mg Plus Docetaxel 75 mg/m^2: Participants with NSCLC were administered with Feladilimab 80 mg IV infusion Q3W in combination with Docetaxel 75 mg/m^2 IV infusion Q3W.
Period: Overall Study
Arm/Group | Docetaxel 75 mg/m^2 | Feladilimab 80 mg Plus Docetaxel 75 mg/m^2
Started | 35 | 70
Completed | 0 | 0
Not Completed | 35 | 70
Not completed — Death | 25 | 62
Not completed — Site Closed | 6 | 6
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Docetaxel 75 mg/m^2 | Feladilimab 80 mg Plus Docetaxel 75 mg/m^2 | Total
Number analyzed (Participants) | 35 | 70 | 105
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.6 (10.48) | 64.4 (9.11) | 63.8 (9.57)
Age, Customized [Count of Participants; unit: Participants]
  18-64 | 22 | 31 | 53
  65-74 | 7 | 28 | 35
  75-84 | 5 | 11 | 16
  >=85 | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 17 | 25
  Male | 27 | 53 | 80
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 35 | 67 | 102
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  Canada | 3 | 0 | 3
  South Korea | 4 | 5 | 9
  Netherlands | 0 | 3 | 3
  Sweden | 0 | 2 | 2
  Romania | 2 | 9 | 11
  United States | 5 | 7 | 12
  Poland | 1 | 3 | 4
  Italy | 4 | 7 | 11
  France | 6 | 9 | 15
  Germany | 3 | 7 | 10
  Spain | 4 | 13 | 17
  Russia | 3 | 5 | 8

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Overall survival was calculated as time from randomization to death. Confidence Intervals estimated using the Brookmeyer Crowley method.
Time Frame: Up to 2 years
Population: Intent To Treat population (ITT) included all participants who were randomized to treatment regardless of whether the participants actually received study treatment.
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Docetaxel 75 mg/m^2: Participants with NSCLC were administered with Docetaxel 75 milligram per meter square (mg/m^2) monotherapy as intravenous (IV) infusion Q3W.
Arm/Group | Docetaxel 75 mg/m^2 | Feladilimab 80 mg Plus Docetaxel 75 mg/m^2
Number analyzed (Participants) | 35 | 70
Months | 8.2 [4.5 to 16.1] | 7.8 [4.7 to 10.8]

2. Secondary Outcome: Kaplan-Meier Estimates of Overall Survival at 12 and 18 Months
Description: Overall survival was defined as the time between date of randomization and death due to any cause. Kaplan-Meier estimates of the percentage of participants who died at each time point was calculated. Confidence Intervals estimated using the Brookmeyer Crowley method.
Time Frame: Month 12 and 18
Population: Intent-To-Treat Population.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Docetaxel 75 mg/m^2 | Feladilimab 80 mg Plus Docetaxel 75 mg/m^2
Number analyzed (Participants) | 35 | 70
Percentage of Participants
  Month 12 | 44 [27 to 60] | 28 [18 to 39]
  Month 18 | 28 [14 to 44] | 18 [10 to 28]

3. Secondary Outcome: Number of Participants With Complete Response (CR), Partial Response (PR), Stable Disease (SD), Progressive Disease (PD) or Not Evaluable
Description: CR, PR, SD and PD will be evaluated as per RECIST version 1.1 criteria. Complete Response (CR) was defined as disappearance of all target and non target lesions and any pathological lymph nodes must be <10 millimeter (mm) in the short axis. Partial Response (PR) was defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as a reference, the baseline sum of the diameters (e.g. percent change from baseline). Stable Disease (SD) was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease. Progressive Disease was defined as at least a 20% increase in the sum of the diameters of target lesions, taking as a reference, the smallest sum of diameters recorded since the treatment started (e.g. percent change from nadir, where nadir is defined as the smallest sum of diameters recorded since treatment start). In addition, the sum must have an absolute increase from nadir of 5mm.
Time Frame: Up to 2 years
Population: Intent-To-Treat Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Docetaxel 75 mg/m^2 | Feladilimab 80 mg Plus Docetaxel 75 mg/m^2
Number analyzed (Participants) | 35 | 70
Participants
  Complete Response | 0 | 0
  Partial Response | 4 | 13
  Stable Disease | 10 | 22
  Progressive Disease | 14 | 23
  Not Evaluable | 7 | 12

4. Secondary Outcome: Kaplan-Meier Estimates of Progression-Free Survival (PFS)
Description: PFS is defined as time from the date of randomization to the date of disease progression as per RECIST v1.1. or death whichever occurs earlier. Progressive Disease was defined as at least a 20% increase in the sum of the diameters of target lesions, taking as a reference, the smallest sum of diameters recorded since the treatment started (e.g. percent change from nadir, where nadir is defined as the smallest sum of diameters recorded since treatment start). In addition, the sum must have an absolute increase from nadir of 5mm. Confidence Intervals estimated using the Brookmeyer Crowley method.
Time Frame: Up to 2 years
Population: Intent to Treat Population. Only those participants with data available at specified data points have been analyzed.
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Feladilimab 80 mg Plus Docetaxel 75 mg/m2: Participants with NSLC were administered with feladilimab 80 mg IV infusion once Q3W in combination with Docetaxel 75 mg/m^2 IV infusion once Q3W.
Arm/Group | Docetaxel 75 mg/m^2 | Feladilimab 80 mg Plus Docetaxel 75 mg/m2
Number analyzed (Participants) | 29 | 62
Months | 3.3 [1.6 to 4.2] | 3.4 [2.6 to 4.3]

5. Secondary Outcome: Objective Response Rate
Description: ORR was calculated as the percentage of participants with a confirmed complete response (CR) or partial response (PR) relative to the total number of participants in the analysis population per response evaluation criteria in solid tumors (RECIST) version (v)1.1. Complete Response (CR) was defined as disappearance of all target and non target lesions and any pathological lymph nodes must be <10 millimeter (mm) in the short axis. Partial Response (PR) was defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as a reference, the baseline sum of the diameters.
Time Frame: Up to 2 years
Population: Intent-To-Treat Population
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Groups:
- Feladilimab 80 mg Plus Docetaxel 75 mg/m2: Participants with NSCLC were administered with feladilimab 80 mg IV infusion Q3W in combination with Docetaxel 75 mg/m^2 IV infusion Q3W.
Arm/Group | Docetaxel 75 mg/m^2 | Feladilimab 80 mg Plus Docetaxel 75 mg/m2
Number analyzed (Participants) | 35 | 70
Percentage of Participants | 11 [3.2 to 26.7] | 19 [10.3 to 29.7]

6. Secondary Outcome: Kaplan-Meier Estimates of Duration of Response (DOR) in Participants With Objective Response
Description: DOR is defined as the time for first documented evidence of CR or PR until disease progression or death, per RECIST 1.1 criteria. Complete Response (CR) was defined as disappearance of all target and non target lesions and any pathological lymph nodes must be <10 millimeter (mm) in the short axis. Partial Response (PR) was defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as a reference, the baseline sum of the diameters. Confidence Intervals estimated using the Brookmeyer Crowley method.
Time Frame: Up to 2 years
Population: Intent To Treat Population. Only participants who achieved Objective Response were evaluated.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Docetaxel 75 mg/m^2 | Feladilimab 80 mg Plus Docetaxel 75 mg/m^2
Number analyzed (Participants) | 4 | 13
Months | 4.8 [2.8 to NA] — Upper limit was not calculated due to insufficient number of participants with events. | 4.3 [2.4 to 8.7]

7. Secondary Outcome: Disease Control Rate (DCR)
Description: DCR is defined as the percentage of participants with a confirmed CR + PR at any time, plus SD =>12 weeks as per RECIST v1.1. Complete Response (CR) was defined as disappearance of all target and non target lesions and any pathological lymph nodes must be <10 millimeter (mm) in the short axis. Partial Response (PR) was defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as a reference, the baseline sum of the diameters (e.g. percent change from baseline). Stable Disease (SD) was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease.
Time Frame: Up to 2 years
Population: Intent-to-Treat Population.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Docetaxel 75 mg/m^2 | Feladilimab 80 mg Plus Docetaxel 75 mg/m^2
Number analyzed (Participants) | 35 | 70
Percentage of Participants | 40 [23.9 to 57.9] | 50 [37.8 to 62.2]

8. Secondary Outcome: Number of Participants With iRECIST Complete Response (iCR), Partial Response (iPR), Unconfirmed Progressive Disease (iUPD), Confirmed Progressive Disease (iCPD), Stable Disease (iSD) or Not Evaluable
Description: Modified RECIST 1.1 for immune-based therapeutics (iRECIST) is based on RECIST v 1.1 but adapted to account for the unique tumor response seen with immunotherapeutic drugs. iRECIST was used to assess tumor response and progression and make treatment decisions. iCR: disappearance of all target lesions; iPR: at least a 30% decrease in the sum of the diameters of target lesions, taking as a reference, the baseline sum of the diameters (e.g. percent change from baseline). iCPD: either 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions; iSD: stable disease in the absence of CR or PD and iUPD: unconfirmed progressive disease when PD is unconfirmed and NE: not evaluable.
Time Frame: Up to 2 years
Population: Intent-To-Treat Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Docetaxel 75 mg/m^2 | Feladilimab 80 mg Plus Docetaxel 75 mg/m^2
Number analyzed (Participants) | 35 | 70
Participants
  iCR | 0 | 0
  iPR | 4 | 13
  iUPD | 11 | 15
  iCPD | 3 | 8
  iSD | 10 | 22
  Not Evaluable | 7 | 12

9. Secondary Outcome: Kaplan-Meier Estimates of iRECIST Progression-free Survival (iPFS)
Description: iPFS is defined as time from the date of randomization to the date of disease progression or death, whichever occurs earlier, per iRECIST criteria. Progressive Disease was defined as at least a 20% increase in the sum of the diameters of target lesions, taking as a reference, the smallest sum of diameters recorded since the treatment started (e.g. percent change from nadir, where nadir is defined as the smallest sum of diameters recorded since treatment start). In addition, the sum must have an absolute increase from nadir of 5mm. Confidence Intervals estimated using the Brookmeyer Crowley method.
Time Frame: Up to 2 years
Population: Intent-to-Treat population. Only those participants with data available at specified data points have been analyzed.
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Feladilimab 80 mg Plus Docetaxel 75 mg/m2: Participants with NSCLC were administered with feladilimab 80 mg IV infusion once Q3W in combination with Docetaxel 75 mg/m^2 IV infusion Q3W.
Arm/Group | Docetaxel 75 mg/m^2 | Feladilimab 80 mg Plus Docetaxel 75 mg/m2
Number analyzed (Participants) | 29 | 62
Months | 3.3 [1.6 to 4.2] | 3.4 [2.6 to 4.3]

10. Secondary Outcome: iRECIST Objective Response Rate (iORR)
Description: iORR is defined as the percentage of participants with a confirmed iCR or iPR at any time per iRECIST criteria. iCR was defined as disappearance of all target and non target lesions and any pathological lymph nodes must be <10 millimeter (mm) in the short axis. iPR was defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as a reference, the baseline sum of the diameters.
Time Frame: Up to 2 years
Population: Intent-to-Treat population.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Docetaxel 75 mg/m^2 | Feladilimab 80 mg Plus Docetaxel 75 mg/m^2
Number analyzed (Participants) | 35 | 70
Percentage of Participants | 11 [3.2 to 26.7] | 19 [10.3 to 29.7]

11. Secondary Outcome: Kaplan-Meier Estimates of iRECIST Duration of Response (iDOR) in Participants With Objective Response
Description: iDOR is defined as the time from first documented evidence of CR or PR until disease progression or death, per iRECIST criteria. iCR was defined as disappearance of all target and non target lesions and any pathological lymph nodes must be <10 millimeter (mm) in the short axis. iPR was defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as a reference, the baseline sum of the diameters. Confidence Intervals estimated using the Brookmeyer Crowley method.
Time Frame: Up to 2 years
Population: Intent-To-Treat Population. Only the participants with Objective Response were evaluated.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Docetaxel 75 mg/m^2 | Feladilimab 80 mg Plus Docetaxel 75 mg/m^2
Number analyzed (Participants) | 4 | 13
Months | 4.8 [2.8 to NA] — Upper limit was not calculated due to insufficient number of participants with events. | 4.3 [2.4 to 8.7]

12. Secondary Outcome: Number of Participants With AEs, Adverse Events of Special Interest (AESI), SAEs and AE/SAEs Leading to Dose Modifications/Delays/Withdrawals
Description: An AE was defined as any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. An SAE was defined as any untoward medical occurrence that, at any dose results in death, is life-threatening, requires in-patient hospitalization or prolongation of existing hospitalization, results in persistent disability/incapacity, is a congenital anomaly/birth defect, any other situation such as important medical events according to medical or scientific judgement. AESI are considered to be Infusion Related Reactions (IRRs) and those of potential immunologic etiology.
Time Frame: Up to 2 years
Population: Safety Population included all the randomized participants who received at least one dose of Standard of Care (SoC), or experimental regimen based on actual treatment received.
Measure: Count of Participants; unit: Participants
Arm/Group | Docetaxel 75 mg/m^2 | Feladilimab 80 mg Plus Docetaxel 75 mg/m^2
Number analyzed (Participants) | 34 | 70
Participants
  AEs | 34 | 70
  AESI | 1 | 4
  SAEs | 16 | 34
  AEs leading to permanent discontinuation of study treatment | 12 | 16
  AEs leading to dose reduction | 7 | 13
  AEs leading to dose interruption/delay | 11 | 24

13. Secondary Outcome: Number of Participants With Maximum Grade Increase in Clinical Chemistry Parameters at Worst Case Post-Baseline
Description: Blood samples were collected for assessment of the clinical chemistry parameters. Laboratory grades were evaluated using the Common Terminology Criteria for Adverse Events (CTCAE v5.0). Grade 1 = Mild AE; Grade 2 = Moderate AE; Grade 3 = Severe AE; Grade 4 = Life-threatening or disabling AE. Number of participants with clinical chemistry results by maximum grade increase (Increase to Grade 3 or Increase to Grade 4) are presented.
Time Frame: Up to 2 years
Population: Safety Population. Only those participants with data available at specified data points have been analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Docetaxel 75 mg/m^2 | Feladilimab 80 mg Plus Docetaxel 75 mg/m^2
Number analyzed (Participants) | 34 | 63
Participants
  Blood bilirubin increased | 0 | 1
  Hypercalcemia: number analyzed (Participants) | 34 | 61
  Hypercalcemia | 0 | 2
  Creatinine increased | 0 | 1

14. Secondary Outcome: Number of Participants With Maximum Grade Increase in Hematology Parameters at Worst Case Post-Baseline
Description: Blood samples were collected for assessment of the hematology parameters. Laboratory grades were evaluated using the Common Terminology Criteria for Adverse Events (CTCAE v5.0). Grade 1 = Mild AE; Grade 2 = Moderate AE; Grade 3 = Severe AE; Grade 4 = Life-threatening or disabling AE. Number of participants with Hematology results by maximum grade increase (Increase to Grade 3 or Increase to Grade 4) are presented.
Time Frame: Up to 2 years
Population: Safety Population. Only those participants with data available at specified data points have been analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Docetaxel 75 mg/m^2 | Feladilimab 80 mg Plus Docetaxel 75 mg/m^2
Number analyzed (Participants) | 34 | 64
Participants
  Anemia | 2 | 5
  Leukocytosis | 0 | 1
  White blood cell decreased | 5 | 11
  Lymphocyte count decreased | 4 | 12
  Neutrophil count decreased | 4 | 13
  Platelet count decreased | 0 | 3

15. Secondary Outcome: Number of Participants With Maximum Grade Increase in Vital Signs (Systolic Blood Pressure and Diastolic Blood Pressure) Parameters at Worst Case Post-Baseline
Description: Blood Pressure was measured after 5 minutes of rest and was taken in the same position throughout the study. Laboratory grades were evaluated using the Common Terminology Criteria for Adverse Events (CTCAE v5.0). Grade 1 = Mild AE; Grade 2 = Moderate AE; Grade 3 = Severe AE. Number of participants with vital signs results by maximum grade increase (Increase to Grade 2 or Increase to Grade 3) are presented.
Time Frame: Up to 2 years
Population: Safety Population. Only those participants with data available at specified time points have been analyzed.
Measure: Count of Participants; unit: Participants
Groups:
- Feladilimab 80 mg Plus Docetaxel 75 mg/m^2: Participants with NSCLC were administered with feladilimab 80 mg IV infusion once Q3W in combination with Docetaxel 75 mg/m^2 IV infusion once Q3W.
Arm/Group | Docetaxel 75 mg/m^2 | Feladilimab 80 mg Plus Docetaxel 75 mg/m^2
Number analyzed (Participants) | 34 | 63
Participants
  Diastolic Blood Pressure | 12 | 26
  Systolic Blood Pressure | 16 | 28

16. Secondary Outcome: Number of Participants With Vital Signs (Temperature) Parameter Results at Worst Case Post-Baseline
Description: Body temperature was measured after 5 minutes of rest. Results are presented in the following categories: Decrease to <=35 Degrees Celsius, Change to Normal or No Change and Increase to >=38 Degrees Celsius.
Time Frame: Up to 2 years
Population: Safety Population. Only those participants with data available at specified data points have been analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Docetaxel 75 mg/m^2 | Feladilimab 80 mg Plus Docetaxel 75 mg/m^2
Number analyzed (Participants) | 34 | 63
Participants
  Decrease to <=35 Degrees Celsius | 0 | 6
  Change to Normal or No Change | 33 | 52
  Increase to >=38 Degrees Celsius | 1 | 5

17. Secondary Outcome: Number of Participants With Vital Signs (Pulse Rate) Parameter Results at Worst Case Post-Baseline
Description: Pulse Rate was measured after 5 minutes of rest. Results are presented in the following categories: Decrease to <50 beats per minute, Change to Normal or No Change and Increase to >120 beats per minute.
Time Frame: Up to 2 years
Population: Safety Population. Only those participants with data available at specified data points have been analyzed.
Measure: Count of Participants; unit: Participants
Groups:
- Docetaxel 75 mg/m^2: Participants with NSLC were administered with Docetaxel 75 milligram per metersquare (mg/m^2) monotherapy as intravenous (IV) infusion once every 3 weeks(Q3W).
- Feladilimab 80 mg Plus Docetaxel 75 mg/m^2: Participants with NSLC were administered with feladilimab 80 mg IV infusion once Q3W in combination with Docetaxel 75 mg/m^2 IV infusion once Q3W.
Arm/Group | Docetaxel 75 mg/m^2 | Feladilimab 80 mg Plus Docetaxel 75 mg/m^2
Number analyzed (Participants) | 34 | 63
Participants
  Decrease to <50 beats per minute | 0 | 0
  Change to Normal or No Change | 32 | 55
  Increase to >120 beats per minute | 2 | 8

18. Secondary Outcome: Minimum Observed Concentration (CmIn) of Feladilimab
Description: Blood samples were collected for assessment of the pharmacokinetic parameters.
Time Frame: Week 1
Population: Pharmacokinetic (PK) population will consist of all participants from the ITT Population from whom a blood sample was obtained and analyzed for PK concentration.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per millimeter (ng/mL)
Arm/Group | Feladilimab 80 mg Plus Docetaxel 75 mg/m^2
Number analyzed (Participants) | 67
nanogram per millimeter (ng/mL) | 6104.6 (91.3)

19. Secondary Outcome: Maximum Observed Concentration (Cmax) of Feladilimab
Description: Blood samples were collected for assessment of the pharmacokinetic parameters.
Time Frame: Week 1, Week 13 and Week 25
Population: Pharmacokinetic population. Only those participants with data available at specified time points have been analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per millimeter (ng/mL)
Arm/Group | Feladilimab 80 mg Plus Docetaxel 75 mg/m^2
Number analyzed (Participants) | 67
nanogram per millimeter (ng/mL)
  Week 1 | 24923.7 (26.7)
  Week 13: number analyzed (Participants) | 34
  Week 13 | 28715.9 (45.4)
  Week 25: number analyzed (Participants) | 15
  Week 25 | 32688.4 (27.4)

20. Secondary Outcome: Maximum Observed Concentration (Cmax) of Docetaxel
Description: Blood samples were collected for assessment of the pharmacokinetic parameters.
Time Frame: Week 1, Week 4, Week 7, Week 10, Week 13, Week 16, Week 19 and Week 22
Population: Pharmacokinetic Population. Only those participants with data available at specified time points have been analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per millimeter (ng/mL)
Arm/Group | Docetaxel 75 mg/m^2 | Feladilimab 80 mg Plus Docetaxel 75 mg/m^2
Number analyzed (Participants) | 30 | 55
nanogram per millimeter (ng/mL)
  Week 1 | 1500.9 (133.5) | 1429.9 (138.7)
  Week 4: number analyzed (Participants) | 29 | 54
  Week 4 | 1587.1 (128.6) | 1399.7 (99.3)
  Week 7: number analyzed (Participants) | 17 | 46
  Week 7 | 846.8 (166.4) | 1036.9 (171.2)
  Week 10: number analyzed (Participants) | 15 | 41
  Week 10 | 1262.9 (155.4) | 1248.4 (118.3)
  Week 13: number analyzed (Participants) | 8 | 32
  Week 13 | 1354.2 (212.1) | 1363.4 (137.8)
  Week 16: number analyzed (Participants) | 6 | 32
  Week 16 | 1095.3 (114.3) | 1381.9 (114.0)
  Week 19: number analyzed (Participants) | 5 | 15
  Week 19 | 759.0 (74.0) | 1765.7 (95.1)
  Week 22: number analyzed (Participants) | 3 | 10
  Week 22 | 535.5 (10.9) | 2430.7 (73.3)

21. Secondary Outcome: Number of Participants With Positive Anti-drug Antibodies (ADA) Against Docetaxel
Time Frame: Up to 2 years
Population: Data was not collected.
Arm/Group | Docetaxel 75 mg/m^2 | Feladilimab 80 mg Plus Docetaxel 75 mg/m^2
Number analyzed (Participants) | 0 | 0

22. Secondary Outcome: Number of Participants With Positive ADA Against Feladilimab
Time Frame: Week 1, 4, 7, 10, 13, 16, 19, 22, 25, 37, 49, 61 and 73
Population: Safety population. Only those participants with data available at specified time points have been analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Feladilimab 80 mg Plus Docetaxel 75 mg/m^2
Number analyzed (Participants) | 69
Participants
  Week 1 | 1
  Week 4: number analyzed (Participants) | 59
  Week 4 | 8
  Week 7: number analyzed (Participants) | 50
  Week 7 | 4
  Week 10: number analyzed (Participants) | 45
  Week 10 | 2
  Week 13: number analyzed (Participants) | 36
  Week 13 | 2
  Week 16: number analyzed (Participants) | 32
  Week 16 | 1
  Week 19: number analyzed (Participants) | 23
  Week 19 | 2
  Week 22: number analyzed (Participants) | 19
  Week 22 | 0
  Week 25: number analyzed (Participants) | 17
  Week 25 | 0
  Week 37: number analyzed (Participants) | 11
  Week 37 | 0
  Week 49: number analyzed (Participants) | 3
  Week 49 | 0
  Week 61: number analyzed (Participants) | 4
  Week 61 | 0
  Week 73: number analyzed (Participants) | 1
  Week 73 | 0

ADVERSE EVENTS:
Time Frame: All cause mortality, non-SAEs and SAEs were collected up to 2 years.
Description: Safety population included all randomized participants who received at least one dose of SoC or experimental regimen based on actual treatment received.
Groups:
- Docetaxel 75 mg/m^2: Participants with NSLC were administered with Docetaxel 75 milligram per meter square (mg/m^2) monotherapy as intravenous (IV) infusion once every 3 weeks (Q3W).
- Feladilimab 80 mg Plus Docetaxel 75 mg/m^2: Participants with NSLC were administered with feladilimab 80 mg IV infusion once Q3W in combination with Docetaxel 75 mg/m^2 IV infusion Q3W.
Arm/Group | Docetaxel 75 mg/m^2 | Feladilimab 80 mg Plus Docetaxel 75 mg/m^2
All-Cause Mortality (participants affected / at risk) | 25/34 | 62/70
Serious Adverse Events (participants affected / at risk) | 16/34 | 34/70
Other Adverse Events (participants affected / at risk) | 31/34 | 66/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Docetaxel 75 mg/m^2 (N=34) | Feladilimab 80 mg Plus Docetaxel 75 mg/m^2 (N=70)
Pneumonia (Infections and infestations) | 6 (7) | 7 (7)
COVID-19 (Infections and infestations) | 0 (0) | 2 (2)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Diarrhoea infectious (Infections and infestations) | 1 (1) | 0 (0)
Lung abscess (Infections and infestations) | 1 (1) | 0 (0)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia mycoplasmal (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 (3) | 4 (4)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Acute respiratory distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Asthenia (General disorders) | 0 (0) | 2 (2)
Chest pain (General disorders) | 0 (0) | 1 (3)
Fatigue (General disorders) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (1)
Performance status decreased (General disorders) | 0 (0) | 1 (2)
Sudden death (General disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Gastric ulcer perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1)
Cardiopulmonary failure (Cardiac disorders) | 0 (0) | 1 (1)
Right ventricular failure (Cardiac disorders) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Troponin increased (Investigations) | 0 (0) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Docetaxel 75 mg/m^2 (N=34) | Feladilimab 80 mg Plus Docetaxel 75 mg/m^2 (N=70)
Asthenia (General disorders) | 10 (11) | 22 (27)
Fatigue (General disorders) | 5 (5) | 17 (22)
Pyrexia (General disorders) | 6 (8) | 12 (14)
Chest pain (General disorders) | 2 (2) | 7 (7)
Mucosal inflammation (General disorders) | 3 (5) | 4 (5)
Oedema peripheral (General disorders) | 1 (1) | 5 (5)
Pain (General disorders) | 1 (2) | 4 (4)
Nausea (Gastrointestinal disorders) | 6 (9) | 26 (45)
Diarrhoea (Gastrointestinal disorders) | 8 (12) | 16 (20)
Constipation (Gastrointestinal disorders) | 2 (2) | 13 (16)
Stomatitis (Gastrointestinal disorders) | 3 (3) | 5 (7)
Vomiting (Gastrointestinal disorders) | 3 (3) | 5 (6)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 4 (4)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 23 (25)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 14 (14)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (5)
Anaemia (Blood and lymphatic system disorders) | 7 (9) | 24 (31)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 12 (16)
Alopecia (Skin and subcutaneous tissue disorders) | 7 (7) | 20 (20)
Nail disorder (Skin and subcutaneous tissue disorders) | 2 (2) | 5 (5)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 7 (7)
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 4 (4)
Weight decreased (Investigations) | 3 (3) | 6 (6)
Blood alkaline phosphatase increased (Investigations) | 2 (2) | 5 (5)
Neutrophil count decreased (Investigations) | 2 (2) | 5 (9)
Alanine aminotransferase increased (Investigations) | 3 (3) | 3 (5)
Blood creatinine increased (Investigations) | 1 (1) | 5 (7)
Blood lactate dehydrogenase increased (Investigations) | 1 (1) | 4 (5)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 2 (2)
White blood cell count decreased (Investigations) | 0 (0) | 4 (10)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 10 (13)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (5) | 7 (7)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 2 (2)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (4)
Paraesthesia (Nervous system disorders) | 3 (3) | 9 (11)
Neuropathy peripheral (Nervous system disorders) | 3 (4) | 5 (5)
Dizziness (Nervous system disorders) | 2 (2) | 4 (4)
Headache (Nervous system disorders) | 2 (2) | 4 (4)
Decreased appetite (Metabolism and nutrition disorders) | 4 (4) | 19 (20)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 5 (5)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Respiratory tract infection (Infections and infestations) | 1 (1) | 5 (5)
Oral candidiasis (Infections and infestations) | 3 (3) | 2 (2)
Urinary tract infection (Infections and infestations) | 1 (1) | 4 (4)
Lacrimation increased (Eye disorders) | 2 (2) | 4 (4)
Insomnia (Psychiatric disorders) | 2 (2) | 4 (4)
Dysuria (Renal and urinary disorders) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2022-05-23): https://cdn.clinicaltrials.gov/large-docs/08/NCT05553808/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-08): https://cdn.clinicaltrials.gov/large-docs/08/NCT05553808/SAP_001.pdf